CLINICAL TRIAL: NCT04830657
Title: The Effect of Reiki on Fatigue and Comfort in Hemodialysis Patients
Brief Title: The Effect of Reiki on Fatigue and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Melek Yesil Bayulgen, Prelector- The Effect of Reiki on Fatigue and Comfort in Hemodialysis Patients, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin Univer
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Hemodialysis; Fatigue
Keywords: Hemodialysis; Reiki; Fatigue; General Comfort; Nursing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial, single masking
Who Masked: Participant
Masking Description: Two groups (n = 31) will be determined by randomization created in computer environment by an independent researcher who is not involved in the study, and patients will be assigned to groups A or B created in computer environment. In determining the groups, lots were made with coins and group A was determined as the control group and group B as the remote reiki group. The information showing that the patients included in the study sample were assigned to the A and B groups according to the randomization table was put in an opaque envelope. This envelope will be kept by the coordinator researcher (MG) and when the researcher (MYB), who has a certificate of reiki application, goes to the patient for the application, he will fill in the "Informed Consent Form" and open the envelope to find out which group the patient is in. If the reiki group far from weakness comes out, the questionnaires will be filled out after verbal consent is obtained from the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distant reiki group (Experimental): The application will be carried out by the researcher who has received level 2 reiki training. Reiki energy will be sent to the individuals who have undergone hemodialysis with the intention of healing. The Reiki practitioner is enabled to send the Reiki remotely in a quiet and lonely room. The practitioner moves to the right side of the individual, imagining as if he is next to the individual, and his aura (the energy that exists around the body) is corrected 3 times from above and from the head to the feet. The practitioner's hands are held side by side. Starting from the beginning of the application, reiki energy is sent to the 7 main chakras in an average of 3 minutes, from top to bottom. Each session is approximately 21-25 minutes. After the session, the chakra equalization process is applied to help the frequencies of the chakras to work in harmony with each other. 15 minutes in total. Balancing is done.
  Interventions: Other: Distant reiki
- Control (Other): Patients will receive routine treatment in accordance with the institution policy without any intervention in the control group.
  Interventions: Other: Distant reiki

INTERVENTIONS:
Other: Distant reiki — In order to determine the sample size of the study, it is planned to study with a total of 62 patients, including at least 31 patients in each group, in the power analysis based on the statistics of the statistician and previous studies. The remote reiki group will be given remote reiki 3 times a week for 4 weeks by the researcher who has a reiki application certificate. Remote reiki sessions will be performed by the reiki practitioner the night before the hemodialysis day of the patient, and the session duration will take approximately 36-40 minutes. After the individuals receive 12 sessions of remote reiki (1 month later), the questionnaire will be filled in for the second measurement. In order to determine whether reiki has an effect in the long term, 4 weeks (1 month) after the second measurement, the questionnaire for the third measurement will be completed and the research will be completed.

SUMMARY:
This study is a single blind, randomized parallel controlled experimental study planned to determine the effect of distant reiki, which is one of the non-pharmacological methods, on fatigue and comfort level in hemodialysis patients. The hypothesis of the study is that distant reiki increases patients comfort and reduces fatigue.

DETAILED DESCRIPTION:
Methods: In order to determine the sample size of the study, before starting the research, power analysis was performed by taking the information of the statistician and previous studies as a reference in order to determine the number of patients to be included in the reiki and control groups. As a result of the analysis performed by taking effect size 0.35, type 1 error 0.05, power 0.80 and correlation between repeated measurements 0.50, it is planned to study with a total of 46 patients, including at least 31 patients in each group. The remote reiki group will be given remote reiki 3 times a week for 4 weeks by the researcher who has a reiki application certificate. Remote reiki sessions will be performed by the reiki practitioner the night before the hemodialysis day of the patient, and the session duration will take approximately 36-40 minutes. After the individuals receive 12 sessions of remote reiki (1 month later), the questionnaire will be filled in for the second measurement. In order to determine whether reiki has an effect in the long term, 4 weeks (1 month) after the second measurement, the questionnaire for the third measurement will be completed and the research will be completed. Patients will receive routine treatment in accordance with the institution policy without any intervention in the control group. The control group will be filled in the questionnaire after the first measurement, in the 4th (1st month) and 8th (2nd month) weeks. At the end of the study, remote reiki sessions will be applied by the researcher, since the patients in the control group have equal ethical rights. The primary expected result of the study is the effect of distant reiki on fatigue in hemodialysis patients. The second expected result of the study is to determine the effect of distant reiki on comfort.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* In patients over the age of 65, the Standardized Mini Mental Test (SMMT) score is 26 and above,
* Having hemodialysis three days / times a week for 6 months or longer with the diagnosis of chronic renal failure,
* Can speak and understand Turkish,
* General condition is good and comfortable (whose life findings are within normal limits)
* Do not have any problem that prevents cognitive, affective and verbal communication,
* Do not use any sedative drugs,
* Do not have any psychiatric illness,
* Those who sign the informed consent form will be included in the sample.

Exclusion Criteria:

* - who do not agree to participate in the study,
* younger than 18,
* In patients over 65 years of age, whose SMMT value is below 24 points
* Patients undergoing hemodialysis without a diagnosis of chronic renal failure,
* Receiving hemodialysis treatment for less than 6 months and once or twice a week,
* Can't speak Turkish,
* General condition unstable (shortness of breath, arrhythmia, fluctuations in blood pressure),
* Diagnosed with anxiety, panic attack and using medication for anxiety,
* Using any sedative medication,
* Have any problem that prevents cognitive, affective and verbal communication,
* Any psychiatric illness,
* Those who do not sign the informed volunteer consent form will not be included in the study.

Study termination criteria:

* Who want to leave the research,
* Changing institution / province,
* If the patient dies, the study will be terminated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Fatigue evaluated using the Fatigue Intensity Index | Change from before implementation, 4th week and 8th week of practice
  The Fatigue Severity Scale will be used to measure the severity of fatigue. The Turkish validity and reliability of the scale, which was developed by Krupp et al in 1989, was carried out in 2007 by Armutlu et al. Each item is scored between 1 and 7 (1 = strongly disagree, 7 = totally agree) in the scale consisting of 9 items that can be applied by individuals in a simple way. The total score range of the scale is 9-63. The total score is calculated by taking the average of 9 items. Accordingly, the lowest average score to be obtained is 1, and the highest average score is 7. The cut-off value was set at 4 and above to diagnose pathological fatigue. The lower the total score, the less fatigue.

SECONDARY OUTCOMES:
Comfort evaluated using the General Comfort Scale | Change from before implementation, 4th week and 8th week of practice
  The Turkish validity and reliability of the scale, which was developed by Kolcaba in 2006, was carried out by Kuğuoğlu and Karabacak in 2008. The scale is 4-point Likert type with 48 items. Comfort theory includes the sub-dimensions of relaxation (9 items), relaxation (9 items) and coping with problems (10 items). There are negative and positive items in the scale. Reverse coding process is applied for negative items, and the lowest total score obtained from the scale is 48 and the highest total score is 192. The mean score of the scale is calculated by dividing the total score obtained from the scale by the number of items. 1 point from the questionnaire indicates low comfort and 4 points indicate high comfort. While Cronbach's alpha reliability coefficient was 0.88 in the reliability study conducted by Kolcaba, it was calculated as 0.85 in the study of Kuğuoğlu and Karabacak who conducted the Turkish validity and reliability study.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No